CLINICAL TRIAL: NCT03049995
Title: The International Stress Echo Study in Ischemic and Non-ischemic Heart Disease
Brief Title: Stress Echo 2020 - The International Stress Echo Study
Acronym: SE2020
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fatebenefratelli Hospital (Other)
Collaborators: Institute of Clinical Physiology, CNR, Pisa,Italy (Unknown); Salerno Hospital, Italy (Unknown); Monaldi Hospital, Napoli, Italy (Unknown); University of Pisa (Other); San Luca Hospital, Lucca, Italy (Unknown); Careggi Hospital (Other); Federico II University (Other); San Carlo Public Hospital, Potenza, Italy (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Ospedale dell'Angelo, Venezia-Mestre (Other); University of Parma (Other); Hospital Clinics, Trieste, Italy (Unknown); Federal University of Rio Grande do Sul (Other); Hospital San José, Criciuma, Brasil (Unknown); Hospital San Vicente de Paulo, Passo Fundo, Brasil (Unknown); University of Belgrade (Other); University of Szeged, Hungary (Unknown); Elisabeth Hospital, Hodmezovasarhely, Hungary (Unknown); Sandro Pertini Hospital, Rome, Italy (Unknown); Hospital Clinics, Bari, Italy (Unknown); Ospedale Nottola, Siena, Italy (Unknown); University of Catania, Italy (Unknown); Medika Cardiocenter, Saint Petersburg, Russian Federation (Unknown); Acibadem City Clinic Tokuda Hospital (Other); Investigaciones Medicas, Buenos Aires, Argentina (Unknown); Tomsk National Research Scientific Centre of Russian Academy of Sciences, Tomsk, Russian Federation (Unknown); Instituto Nacional de Cardiología Mexico City, Mexico (Unknown); Hamad Medical Corporation, Heart Hospital -Doha-Qatar (Unknown)
Responsible Party: Sponsor
Other Study IDs: FBF001
Record Dates: First submitted 2017-02-02; First posted 2017-02-10 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Heart Failure; Hypertrophic Cardiomyopathy; Aortic Valve Disease; Athletes Heart; Tetralogy of Fallot; Pulmonary Arterial Hypertension
Keywords: effectiveness; imaging; prognosis; stress echocardiography
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Cardiomyopathy, Hypertrophic; Aortic Valve Disease; Tetralogy of Fallot; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and saliva will be collected in patients of "GENES"protocol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- CHEF:Cardiac Resynchronization therapy Forecast: Patients evaluated prior to cardiac resynchronization therapy (CRT), with class I, IIa or IIb for CRT according to ESC 2016 guidelines, and with ejection fraction ≤ 35% and QRS duration ≥ 130 ms. Contractile reserve will be assessed through variations in Wall Motion Score Index and with more advanced parameters such as left ventricular elastance reserve, as the peak stress/baseline ratio of end - systolic pressure/ end-systolic volume (Left ventricular contractile reserve SE). All patients will be followed-up with resting echocardiographic examination to assess left ventricular remodelling and recovery of function. A sample size of 277 patients is required and about the same number is required to predict the response to medical therapy in patients eventually not undergoing CRT (4).
  Interventions: Procedure: Left ventricular contractile reserve SE
- BHEF: B-lines in HEart Failure: B- lines are a semiquantitative sign of extravascular lung water present in 1 out of 3 HF patients at rest and in 1 out of 2 during stress, and potentially useful for refining prognostic stratification and titrating diuretic therapy in these patients. We will enroll patients referred to SE with known or suspected HF, with either reduced or preserved ejection fraction. B-lines will be detected using the B-lines SE intervention. A sample size of about 2500 patients is required if the effect on mortality is evaluated.
  Interventions: Procedure: B-lines SE
- SEHCA: SE in Hypertrophic Cardiomyopathy: Current guidelines recommend SE in hypertrophic cardiomyopathy (HC) solely for evaluation of left ventricular outflow tract obstruction. Large-scale registry data show that SE positivity for ischemic criteria rather than provocable gradients predict adverse outcome in HC. Low-to-intermediate risk symptomatic or asymptomatic HC patients will undergo exercise SE with assessment at each stage and during recovery of wall motion, mitral insufficiency, left ventricular outflow tract gradient (in orthostatic position)(following specific SE protocol), E/e', B-lines and, if feasible, coronary flow velocity reserve. A sample size of about 250 patients is required.
  Interventions: Procedure: B-lines SE; Procedure: Left ventricular outflow tract gradient SE
- SEDIA: SE in Diastolic Heart failure: Patients with suspected diastolic heart failure according to guidelines (3) will be selected (1).The diastolic assessment should be included into all exercise SE tests by measuring standard Doppler-derived mitral inflow velocity, pulsed Tissue Doppler of mitral annulus, and retrograde tricuspid gradient of tricuspid regurgitation as well as diastolic left ventricular volume index and B-lines (to provide a direct imaging of extra-vascular lung water accumulation as a direct cause of dyspnea). The test is considered positive for diastolic dysfunction when all of the following three conditions are met during exercise: average E/e' > 14 or septal E/e' ratio > 15, peak tricuspid regurgitant jet velocity >2.8 m/sec and septal e' velocity < 7 cm/s. A sample size of about 250 patients is required.
  Interventions: Procedure: Diastolic function SE
- SETA: SE in Transcatheter Aortic Valve implantation: Transcatheter Aortic Valve Implantation is an extraordinarily effective novel technology, and its short and long term morbidity and mortality remains significant. Patients with previous (from 6 months to 10 years) surgical or Transcatheter Aortic Valve Implantation capable of exercising will be enrolled and studied with semisupine SE. The full quantitative evaluation of mitral regurgitation and aortic stenosis will be performed. A sample size of about 100 patients is required to detect a significant stress-induced increase in mitral regurgitation severity. For the prognostic analysis 250 patients with 3 years follow-up are required.
  Interventions: Procedure: Mitral regurgitation SE
- SEO: SE in Outdoor in Extreme conditions: SE can also be performed outdoors, with pocket size or portable instruments, in a setting of ecological stress entirely different from standard indoor testing. The diagnostic target is the early subclinical identification of pulmonary edema. Subjects involved in extreme sporting events (competitive triathlon, marathon, apnea diving etc) or ordinary exercise in extreme environments (trekking at high altitude) will undergo lung ultrasound scan for B-lines before, soon after (within 10 minutes) and (when positive) soon after, later after (6 to 24 h) the acute extreme exercise. A sample size of 80 patients is required to detect a significant stress-induced increase in B-lines in each of the three major study subgroups: high altitude trekkers (n=100); marathon runners (n=80) and apnea divers (n=70).
  Interventions: Procedure: B-lines SE
- SETOF: SE in operated Tetralogy of Fallot: Patients with repaired Tetralogy of Fallot or Fallot-like pathology (double-outlet right ventricle Fallot type, tetralogy of Fallot with pulmonary atresia), evaluated at least 1 year after the last surgical or percutaneous procedure, will be recruited by regional reference centers for congenital heart disease. Additional inclusion criteria are age > 10 years, height > 140 cm, New York Heart Association class I or II. Right ventricular function will be assessed at baseline and peak stress with variations (rest and peak stress) of tricuspid annular plane systolic excursion. A sample size of about 250 patients is required to detect a significant stress-induced increase in tricuspid annular plane systolic excursion.
  Interventions: Procedure: Pulmonary hemodynamics SE
- DOSPAH: Doppler SE in Pulmonary Arterial Hypertension: Patients at risk, borderline, or early established pulmonary hypertension capable of exercising will be recruited by regional reference centers, a physical stress will be performed and the hemodynamic assessment will include the assessment of pulmonary hemodynamics. The primary positivity criteria are the increase in systolic pulmonary artery pressure (> 40 mmHg) and the flow-adjusted variation in pulmonary vascular resistances. A sample size of about 250 patients is required to detect a significant stress-induced hemodynamic changes with a 3 -year follow-up.
  Interventions: Procedure: Pulmonary hemodynamics SE
- DITSE: Diagnosis of CAD by imaging SE: A clear step-up in diagnostic sensitivity (with a modest loss in specificity) and risk stratification capability is obtained with assessment of coronary flow velocity reserve in the left anterior descending coronary artery,left ventricular contractile reserve through changes in left ventricular elastance, and B-lines. "Allcomers" referred to the SE lab with suspected CAD will be evaluated with standard regional wall motion analysis and also - whenever feasible - with left ventricular coronary flow reserve and left ventricular elastance reserve and - when possible- B-lines ("quadruple imaging").A sample size of about 5,000 patients will be required.
  Interventions: Procedure: Left ventricular contractile reserve SE; Procedure: B-lines SE; Procedure: Coronary flow reserve SE
- GENES: Genetic Stress echocardiography: The identification of phenotype-negative and genotype positive carriers of pathologic mutations is an important, still elusive, target. We will initially select 75 patients (25 for each disease) with documented disease and mutant gene. We will enroll 250 first-degree relatives of the initially considered probands, with normal findings at rest and age range preferentially between 10 and 21 years. SE testing will be tailored on the specific question: hypertrophic cardiomyopathy as in protocol 3 (left ventricular outflow tract gradient); pulmonary hypertension as in protocol 8 (pulmonary vascular resistances);dilated cardiomyopathy as in protocol 1 (left ventricular elastance). A sample size of about 80 patients for each disease will be required.
  Interventions: Procedure: Left ventricular contractile reserve SE; Procedure: Left ventricular outflow tract gradient SE; Procedure: Pulmonary hemodynamics SE

INTERVENTIONS:
Procedure: Left ventricular contractile reserve SE — Stress protocols (either physical or pharmacological) will be performed according to recent guidelines recommendations (1,2,3). with special focus on Wall Motion Score Index.
  Groups: CHEF:Cardiac Resynchronization therapy Forecast; DITSE: Diagnosis of CAD by imaging SE; GENES: Genetic Stress echocardiography
Procedure: B-lines SE — SE will be performed with special focus on lung sonography and B-lines score (3,4).B-lines will be scored with the 28-regions antero-lateral chest assessment as previously described at baseline and immediately after stopping exercise. A simplified 8-region scan is also allowed in order to save time without loss of critical information.
  Groups: BHEF: B-lines in HEart Failure; DITSE: Diagnosis of CAD by imaging SE; SEHCA: SE in Hypertrophic Cardiomyopathy; SEO: SE in Outdoor in Extreme conditions
Procedure: Left ventricular outflow tract gradient SE — SE will be performed with special focus on left ventricular outflow tract obstruction (3,4).
  Groups: GENES: Genetic Stress echocardiography; SEHCA: SE in Hypertrophic Cardiomyopathy
Procedure: Diastolic function SE — SE will be performed with special focus on E/e', pulmonary artery systolic pressure, B-lines and left ventricular end-diastolic volume (3,4).
  Groups: SEDIA: SE in Diastolic Heart failure
Procedure: Mitral regurgitation SE — SE will be performed with special focus on mitral regurgitation and aortic valve gradients assessment (3,4).
  Groups: SETA: SE in Transcatheter Aortic Valve implantation
Procedure: Pulmonary hemodynamics SE — SE will be performed with special focus on pulmonary artery systolic pressure and pulmonary artery hemodynamics.
  Groups: DOSPAH: Doppler SE in Pulmonary Arterial Hypertension; GENES: Genetic Stress echocardiography; SETOF: SE in operated Tetralogy of Fallot
Procedure: Coronary flow reserve SE — SE will be performed with special focus on regional wall motion + coronary artery flow velocity reserve.
  Groups: DITSE: Diagnosis of CAD by imaging SE

SUMMARY:
Background: Stress echocardiography (SE) has an established role in evidence-based guidelines, but recently the breadth and variety of applications has extended well beyond coronary artery disease (CAD). Purpose: To establish a prospective research study of SE applications, in and beyond CAD, also considering a variety of signs in addition to regional wall motion abnormalities. Methods: In a prospective, multicenter, international, observational study design, > 100 certified high-volume SE labs will be networked with an organized system of clinical, laboratory and imaging data collection at the time of physical or pharmacological SE, with structured follow-up information. The study is endorsed by the Italian Society of Echocardiography and organized in 10 subprojects focusing on: contractile reserve for prediction of cardiac resynchronization or medical therapy response; stress B-lines in heart failure; hypertrophic cardiomyopathy; heart failure with preserved ejection fraction; mitral regurgitation after either transcatheter or surgical aortic valve replacement; outdoor SE in extreme physiology; right ventricular contractile reserve in repaired tetralogy of Fallot; suspected or initial pulmonary arterial hypertension; coronary flow velocity, left ventricular elastance reserve and B-lines in known or suspected CAD; identification of subclinical familial disease in phenotype-negative healthy relatives of inherited disease (such as hypertrophic cardiomyopathy). Expected Results:To collect about 10,000 patients over a 5-year period (2016-2020), with sample sizes ranging from 5,000 for known or suspected CAD to around 250 for hypertrophic cardiomyopathy or repaired Fallot. This data base will allow to investigate technical questions such as feasibility and reproducibility of various SE parameters and to assess their prognostic value in different clinical scenarios. Conclusions: The study will create the cultural, informatic and scientific infrastructure connecting high-volume, accredited SE labs, to obtain original safety, feasibility, and outcome data in evidence-poor diagnostic fields, also outside the established core application of SE in CAD based on regional wall motion abnormalities. The study will standardize procedures, validate emerging signs, and integrate the new information with established knowledge, helping to build a next-generation SE lab without inner walls.

DETAILED DESCRIPTION:
In a prospective, multicenter, international, observational study design, > 100 SE labs will be networked with systematic clinical, laboratory and imaging data collection at the time of SE and with structured follow-up information at least at 6 months and 1 year, up to 3 years for specific protocols. For all the groups the primary aim is to evaluate the feasibility of several indices of SE in the evaluation of patients with known or suspected specific disease (1,2,3). The secondary aim is to assess the value of each of these parameters in predicting the functional impairment. The tertiary aim is to assess the prognostic value of SE indices for prognostic stratification of the disease in the medium-long-term.

The study theater is the international network of cardiology SE laboratories, and the study is endorsed and promoted by the Italian Society of Echocardiography. The starting point of the recruitment phase was a recent electronic survey by the Italian Society of Echocardiography, in 2015 censoring 134 laboratories with moderate- (>100/year) to high- (>400/year) volume SE activities, which were precisely interrogated for interest in participation to SE2020. The recruitment plan forecasts 500 patients by the end of 2016, with doubling of the rate of enrollment in subsequent years, in parallel with the increasing number of recruiting labs fulfilling quality control criteria, reaching the target number of 100 at the end of the 5-year schedule (4).

Data collection Stress protocols are harmonized according to recent European and North-American scientific societies' guidelines, with semi-supine exercise recommended and pharmacological stress dosages up to 40 mcg/kg/min for dobutamine, up to 0.84 mg/kg in 6 min for dipyridamole, and up to a 4-min step of 200 microg/kg/min for adenosine. With dobutamine, atropine (up to 1 mg) can be administered in patients with suspected CAD (protocol 9), and it is associated with a higher rate of complications in those with a history of neuropsychiatric symptoms, reduced left ventricular function, or small body habitus. The maximal allowed dobutamine dose is 20 mcg/kg/min in patients with aortic stenosis, in whom higher doses are less safe and probably unnecessary (3). All laboratories will share a standardized case report form coded in a database format to facilitate retrieval and communication. For applications outside CAD and for CAD testing with vasodilator stress, no atropine is given on top of pharmacological stress. Although data collection with a dedicated project-specific case report form is allowed, we encourage implementing a dedicated, free ad-hoc system for data storage and reporting developed at the National Research Council, Institute of Clinical Physiology. The software provides a suitable informatics infrastructure for the SE 2020 Italian multicenter study, with an intuitive graphic interface, eye-catching graphic format and convenient reporting option. It could represent the trade-off between the comprehensive information required by scientific standards and the smooth workflow priority of busy, high-volume, clinically-driven activities. The software was developed and tested in Italian and the translation of the last release in other languages (English, Portuguese and Serbian) is currently in progress.

Data analysis Data will be expressed as mean ± standard deviation (normally distributed data, such as wall motion score index), median and inter-quartile (25th, 75th) range (non-normally distributed data, such as B-lines) or per cent frequency (categorical data, such as presence or absence of severe mitral regurgitation), with absolute numbers. One-sample comparisons will be performed using Wilcoxon test, and the chi-squared test without Fisher's correction for categorical data. Event rates will be estimated with Kaplan-Meier curves and compared by the log-rank test. Univariable analyses by Cox proportional hazards models will be performed to assess the association between each candidate variable and outcome. All variables with P <0.20 by univariable analysis will be considered as candidate variables for the multivariable analyses. Goodness of fit of the models will be based on C-statistics and its variants, adjusting for optimism using bootstrap replications (at least 1000). A receiver operating characteristic analysis will be used to obtain the best prognostic predictor for the individual SE variables. We will also analyze the data according to a clinically guided stepwise procedure, where the variables were included in the model in the same order in which they are actually considered by the cardiologist. Statistical significance will be set at p<0.05.

Quality control

It is well-known that the diagnostic performance of SE is closely related to the level of expertise of the cardiologist-echocardiographer performing the test, since the evaluation of regional wall motion is subjective and qualitative, with considerable variability even among experienced centers of undisputed reputation (1). The reproducibility and accuracy of wall motion reading can be substantially increased with limited training (2) and through development of conservative, pre-specified reading criteria (4). Therefore, quality control of the diagnostic performance in the various laboratories is a must in order to enter meaningful information in the data bank. The burden of quality control is on the hub center of the principal investigator of each subproject, where various spoke centers may converge. For the general project, the hub center for regional wall motion analysis is Pisa-CNR, in coordination with the principal investigator. There are five different levels of quality control, with increasing levels of complexity:

1. Level 1, pre-requisite: a volume activity of the lab of at least 100 SE tests per year, which is the requirement for credentialing of SE activity by scientific societies
2. Level 2, spoke centers read hub SE images, consisting in 20 selected studies for regional wall motion analysis. The concordance requires identification of test negativity/positivity and, in positive tests, the correct localization of the ischemic zone. For each test, a multiple choice 6-answer test is given. The criterion of ≥ 90% concordance (at least 18 out of 20 studies) is required, as previously described for first-generation SE multicenter studies (4).
3. Level 3, hub centers read spoke centers studies, consisting in 20 any-quality consecutive studies recorded by the spoke center. The criterion of ≥ 80% concordance (at least 16 out of 20 studies) is required, as previously described for first-generation SE multicenter studies (4).
4. Level 4, core lab reading. All centers should grant full access to images of SE studies entered in the data bank for audit or reading by core lab laboratory, which is the standard for specific subprojects such as number 10 for genetic SE, when every effort needs to be made to minimize variability and a single reader will analyze all studies acquired by different centers, as required by recommendations for small-to-medium sample studies, when resources allow (4).
5. Level 5, specific protocols quality control. Although the SE quality control has proved to work well for regional wall motion analysis, novel SE applications involve different parameters, methodology of acquisition and reading criteria. Therefore, for each subproject, a web-based training session and quality control is organized by the specific hub center and principal investigator to assure consistency of data (4). The principal investigator of each subproject will prepare a set of 20 studies with rest-stress images. For each test, a multiple choice 6-answers test is given (only 1 correct). The criterion of ≥90% concordance (at least 18 out of 20 studies) is required. The specific signs tested for certification are: end-diastolic and end-systolic volume changes (protocol 1); B-lines (protocol 2, 4, 6 and 9); left ventricular outflow tract gradient (protocol 3 and 10); E/e' (protocol 4); mitral regurgitation quantitative assessment (protocol 5); aortic stenosis quantitative assessment (protocol 5); right ventricular function (protocol 7); systolic pulmonary artery pressure measurements during stress (protocol 8); coronary flow velocity reserve (protocol 9); left ventricular elastance (protocol 9); global longitudinal strain (protocol 4 and 10).

This study is also intended as a special level of voluntary accreditation and expertise in the specific field of interest, well above the volume activity criteria requested by guidelines. The accreditation process is run and certified by the Italian scientific society of echocardiography strictly following criteria and procedures of the European association of cardiovascular imaging to ensure standardization and independence of the process. When not otherwise specified, resting and SE measurements are performed according to the latest joint recommendations of European and North-American societies (4).

Overall study design We will collect the experience of Italian, Brazilian, Hungarian and Serbian SE labs over the 5-year period from 2016 to 2020. In this broader framework, 10 sub-projects will address specific patients' subsets. The target population ranges from 250-patient samples for protocols focused on specific diseases (such as protocol 7 in repaired tetralogy of Fallot) to 2,500 for protocols on heart failure (number 2) to 5,000 to all-comers with known or suspected CAD tested with novel indices (number 9).

Different study projects will cover the entire spectrum of disease, age and clinical status of current patients. The recruited participants are "the wellest of the well" (super-fit athletes entering project 6), the "worried well" (young first-degree relatives of patients with hypertrophic cardiomyopathy or familiar forms of dilated cardiomyopathy or pulmonary arterial hypertension, in project 10), the "suspected sick" (for instance patients with suspected diastolic heart failure or CAD as in projects 4 and 9), up to the sickest of the sick (for instance, patients with advanced heart failure or valvular heart disease entering projects 1, 2 and 5). Some degree of overlap is unavoidably present for some projects, for instance with subjects eligible for project 2 who are also recruitable for project 1 (if they undergo cardiac resynchronization therapy) or for project 5 (if they have heart failure with preserved ejection fraction). Over time, patients may move from one project to another: for instance, first-degree relatives of hypertrophic cardiomyopathy patients with negative phenotype enrolled in project 10 may subsequently develop overt forms of disease and be enrolled in project 3. All these potential gray-zone situations will be readily identified in individual SE reports.

Although the setting will be mainly the Italian cardiological community, all essential documents will be written in English and we plan to extend the project to other communities with long-standing history of cooperation and experience in multicenter trials. Brazilian, Hungarian and Serbian centers are already recruiting and additional laboratories from other countries are now entering the process of accreditation. The project is curiosity-driven, independent from sponsors, and clinically oriented. However, after the planning and start-up phase, support from public or private funding agencies or industries is possible - provided that it is unrestricted and does not interfere in any way with data collection and analysis.

There is no bonus payment for subject recruitment and subject referral. Enrolled patients are referred to the SE lab for clinically-driven indications. Each patient signs an informed consent form allowing scientific utilization of data, respectful of privacy rights, at the time of testing. The study project was submitted by the coordinating center of the principal investigator on January 31, 2016 and approved in its revised form by the Rome-1 ethical committee on July 20, 2016 (protocol number 1487/Lazio1). Ethics committee approval will be sought by each participating center, as needed.

ELIGIBILITY:
Inclusion criteria shared by all projects are:

* age < 85 years and > 18 years (except for project 7 regarding repaired tetralogy of Fallot and project 10 regarding healthy relatives of patients with familial disease, in which children > 10 years can enter the study after parental consent);
* technically acceptable acoustic window at rest (with at least 14 segments well visualized in at least one projection).

Exclusion criteria shared by all projects are:

* presence of prognosis-limiting comorbidities, such as advanced cancer, reducing life expectancy to < 1 year;
* pregnancy/lactation;
* unwillingness to give informed consent and to enter a regular follow-up program.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Heart Failure patients candidates for cardiac resynchronization therapy.
  2. Patients with known or suspected HF.
  3. Hypertrophic cardiomyopathy.
  4. HF with preserved ejection fraction.
  5. Patients with aortic valve replacement.
  6. Healthy volunteers involved in extreme sporting events (competitive triathlon, marathon, apnea diving etc).
  7. Tetralogy of Fallot operated patients.
  8. At risk borderline, or early established pulmonary hypertension.
  9. Known or suspected CAD.
  10. First degree relatives with familial dilated cardiomyopathy, pulmonary hypertension or hypertrophic cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
all cause death | 5 years
  Death from any cause occurring between 5 years after the time of SE enrollment
cardiac death | 5 years
  Death from cardiac cause occurring between 5 years after the time of SE enrollment
transplantation | 5 years
  Cardiac transplantation occurring between 5 years after the time of SE enrollment

SECONDARY OUTCOMES:
clinical (NYHA class IV) or functional (EF 30>10%) | 5 years
  signs and symptoms consistent with heart failure which required hospitalization between 5 years after the time of SE enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Quirino Ciampi, MD, Principal Investigator — Fatebenefratelli Hospital
Locations (1):
- Fatebenefratelli Hospital, Benevento, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellikka PA, Nagueh SF, Elhendy AA, Kuehl CA, Sawada SG; American Society of Echocardiography. American Society of Echocardiography recommendations for performance, interpretation, and application of stress echocardiography. J Am Soc Echocardiogr. 2007 Sep;20(9):1021-41. doi: 10.1016/j.echo.2007.07.003. No abstract available. PMID 17765820
- [Background] Sicari R, Nihoyannopoulos P, Evangelista A, Kasprzak J, Lancellotti P, Poldermans D, Voigt JU, Zamorano JL; European Association of Echocardiography. Stress Echocardiography Expert Consensus Statement--Executive Summary: European Association of Echocardiography (EAE) (a registered branch of the ESC). Eur Heart J. 2009 Feb;30(3):278-89. doi: 10.1093/eurheartj/ehn492. Epub 2008 Nov 11. No abstract available. PMID 19001473
- [Background] Lancellotti P, Pellikka PA, Budts W, Chaudhry FA, Donal E, Dulgheru R, Edvardsen T, Garbi M, Ha JW, Kane GC, Kreeger J, Mertens L, Pibarot P, Picano E, Ryan T, Tsutsui JM, Varga A. The clinical use of stress echocardiography in non-ischaemic heart disease: recommendations from the European Association of Cardiovascular Imaging and the American Society of Echocardiography. Eur Heart J Cardiovasc Imaging. 2016 Nov;17(11):1191-1229. doi: 10.1093/ehjci/jew190. PMID 27880640
- [Background] Picano E, Ciampi Q, Citro R, D'Andrea A, Scali MC, Cortigiani L, Olivotto I, Mori F, Galderisi M, Costantino MF, Pratali L, Di Salvo G, Bossone E, Ferrara F, Gargani L, Rigo F, Gaibazzi N, Limongelli G, Pacileo G, Andreassi MG, Pinamonti B, Massa L, Torres MA, Miglioranza MH, Daros CB, de Castro E Silva Pretto JL, Beleslin B, Djordjevic-Dikic A, Varga A, Palinkas A, Agoston G, Gregori D, Trambaiolo P, Severino S, Arystan A, Paterni M, Carpeggiani C, Colonna P. Stress echo 2020: the international stress echo study in ischemic and non-ischemic heart disease. Cardiovasc Ultrasound. 2017 Jan 18;15(1):3. doi: 10.1186/s12947-016-0092-1. PMID 28100277
- [Derived] Merli E, Ciampi Q, Scali MC, Zagatina A, Merlo PM, Arbucci R, Daros CB, de Castro E Silva Pretto JL, Amor M, Salame MF, Mosto H, Morrone D, D'Andrea A, Reisenhofer B, Rodriguez-Zanella H, Wierzbowska-Drabik K, Kasprzak JD, Agoston G, Varga A, Lowenstein J, Dodi C, Cortigiani L, Simova I, Samardjieva M, Citro R, Celutkiene J, Re F, Monte I, Gligorova S, Antonini-Canterin F, Pepi M, Carpeggiani C, Pellikka PA, Picano E; Stress Echo 2020 and 2030 study group of the Italian Society of Echocardiography and Cardiovascular Imaging (SIECVI). Pulmonary Congestion During Exercise Stress Echocardiography in Ischemic and Heart Failure Patients. Circ Cardiovasc Imaging. 2022 May;15(5):e013558. doi: 10.1161/CIRCIMAGING.121.013558. Epub 2022 May 17. PMID 35580160
- [Derived] Scali MC, Zagatina A, Ciampi Q, Cortigiani L, D'Andrea A, Daros CB, Zhuravskaya N, Kasprzak JD, Wierzbowska-Drabik K, Luis de Castro E Silva Pretto J, Djordjevic-Dikic A, Beleslin B, Petrovic M, Boskovic N, Tesic M, Monte I, Simova I, Vladova M, Boshchenko A, Vrublevsky A, Citro R, Amor M, Vargas Mieles PE, Arbucci R, Merlo PM, Lowenstein Haber DM, Dodi C, Rigo F, Gligorova S, Dekleva M, Severino S, Lattanzi F, Morrone D, Galderisi M, Torres MAR, Salustri A, Rodriguez-Zanella H, Costantino FM, Varga A, Agoston G, Bossone E, Ferrara F, Gaibazzi N, Celutkiene J, Haberka M, Mori F, D'Alfonso MG, Reisenhofer B, Camarozano AC, Miglioranza MH, Szymczyk E, Wejner-Mik P, Wdowiak-Okrojek K, Preradovic-Kovacevic T, Bombardini T, Ostojic M, Nikolic A, Re F, Barbieri A, Di Salvo G, Merli E, Colonna P, Lorenzoni V, De Nes M, Paterni M, Carpeggiani C, Lowenstein J, Picano E; Stress Echo 2020 Study Group of the Italian Society of Echocardiography and Cardiovascular Imaging. Lung Ultrasound and Pulmonary Congestion During Stress Echocardiography. JACC Cardiovasc Imaging. 2020 Oct;13(10):2085-2095. doi: 10.1016/j.jcmg.2020.04.020. Epub 2020 Jul 15. PMID 32682714